CLINICAL TRIAL: NCT06543667
Title: A Clinical Study for Safety and Efficacy Evaluation of Limbal Stem Cell Derived Exosome (LSC-Exo) Eye Drop for Treatment of Dry Eye Syndrome
Brief Title: Limbal Stem Cell Derived Exosome (LSC-Exo) Eye Drop for Treatment of Dry Eye
Acronym: EXOIUMS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Shoae Hassani, Director, Iran University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRCT20231022059814N1; 1358-06 (Other Grant/Funding Number: Cellule Daru Darman Iranian (Cell Pharma))
Record Dates: First submitted 2024-08-04; First posted 2024-08-09 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-08

CONDITIONS: Dry Eye Syndromes
Keywords: Dry Eye Disease; Sjogren's Syndrome; Chronic Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Limbal Stem Cell Derived Exosome Eye Drop treatment (Experimental): Patients will receive artificial tears for 2 weeks to get the normalized baseline, followed by LSC-Exo eye drop intervention for 3 months.
  Interventions: Biological: Limbal Stem Cell Derived Exosomes Eye Drop

INTERVENTIONS:
Biological: Limbal Stem Cell Derived Exosomes Eye Drop — Patients will receive artificial tears for 2 weeks to get the normalized baseline, followed by LSC-Exo eye drops 0.15 ml/single eye/one time, four times a day for 3 months. The follow-up visit will be 12 weeks since the administration of LSC-Exo eye drops.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Limbal Stem Cells derived Exosomes (LSC-Exo) in alleviation of dry eye symptoms

DETAILED DESCRIPTION:
Dry eye is among the most prevalent chronic conditions in ophthalmology, significantly impacting quality of life and presenting a public health challenge that cannot be overlooked. Current treatment options primarily consist of artificial tear replacement, anti-inflammatory therapies, and local immunosuppressive treatments, which mainly focus on alleviating discomfort and other symptoms associated with the ocular surface. However, with the rapid advancements in regenerative medicine, ophthalmologists are exploring innovative approaches to treat dry eye. Chronic dry eye can result in corneal damage and potential vision loss. Recent studies suggest that therapeutic exosomes delivered as eye drops can enhance the immune microenvironment of the cornea and alter the ocular surface's microenvironment for better outcomes.

Exosomes are membrane vesicles secreted by parental cells, which can mediate the transfer of RNA, protein, DNA and other functional molecules of the parent cell between other cells and regulate the function of target cells. The therapeutic potential of Limbal Stem Cell Exosomes has been studied by our department. We found that LSC-Exo can alleviate the symptoms of dry eye in the animal study. At present, we plan to clarify its efficacy in a clinical research.

The main objective of this study is to evaluate the alleviation of Dry Eye symptoms in patients which are resist to conventional treatment by tear drops. The assessment will be done after LSC-Exo treatment by measuring Ocular Surface Index Score (OSDI), and the second objective include the measurement of inflammatory and pro-inflammatory cytokines in tear of patients, tear secretion amount, tear break time, the areas stained by fluorescent, ocular redness, tear meniscus and best corrected visual acuity.

Approximately 30 patients will be recruited. The treatment group will receive artificial tears for 2 weeks to normalize the baseline, followed by intervention of LSC-Exo 10ug/drop, four times a day for 30 days. The follow-up visit will be 12-weeks and the progression of dry eye will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complaints of burning or itching or feeling of a foreign body in the eye
* Moderate and severe dry eye severity
* Age between 18-70 years

Exclusion Criteria:

* Previous history of eye surgery
* Any disease that suppresses the immune system
* Pregnancy and breastfeeding
* Eyelid abnormalities
* Use of eye drops in the past year except artificial tears and lubricating ointments
* Use of systemic drugs that affect the tear film in last three months
* Use of contact lenses in the last three months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Inflammatory and Pro-inflammatory cytokines changes | 12 weeks
  Dry eye is characterized by ocular surface inflammation. Proinflammatory cytokines IL-1, IL-6, IL-8, TNF-α and IFN-γ are strongly correlated with dry eye markers, leading to ocular surface damage.
Change in Ocular Surface Disease Index (OSDI) | 4, 8 , and 12 weeks
  The OSDI questionnaire contains 12 questions to measure dry eye symptoms. OSDI scores range from 0 to 100. The lower the score, the more alleviation of dry eye symptoms. Compared with the baseline, a reduction of more than 10 points indicates improvement

SECONDARY OUTCOMES:
Tear Secretion Test (Schirmer test) | 4, 8 , and 12 weeks
  A paper strip is placed on the eye under the lower lid for a specified time period. The length of the strip wetted by the tears was measured in millimeters. A positive change from baseline indicates an improvement in each eye.
Tear Film Break-up Time | 4, 8 , and 12 weeks
  Time required for dry spots to appear on the surface of the eye after blinking was measured in seconds. A positive change from baseline indicates improvement in each eye.

CONTACTS AND LOCATIONS:
Locations (1):
- Moheb Kowsar Hospital, Tehran, Iran

REFERENCES:
- [Derived] Randall Harrell C, Djonov V, Volarevic A, Arsenijevic A, Volarevic V. Mesenchymal Stem Cell-Sourced Exosomes as Potentially Novel Remedies for Severe Dry Eye Disease. J Ophthalmol. 2025 Jan 10;2025:5552374. doi: 10.1155/joph/5552374. eCollection 2025. PMID 39839752